CLINICAL TRIAL: NCT03859921
Title: A Randomized Double Blind Controlled Comparison of Oral Dydrogesterone as Luteal Phase Support in Natural Cycle Frozen-thawed Embryo Transfer
Brief Title: Oral Dydrogesterone as Luteal Phase Support in Natural Cycle FET
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW 18-594
Record Dates: First submitted 2019-02-26; First posted 2019-03-01 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-03

CONDITIONS: Subfertility
MeSH Terms: conditions — Infertility | interventions — Dydrogesterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dydrogesterone group (Experimental): Oral dydrogesterone 10mg tds will be given for two weeks from the next day of the LH surge or hCG induced ovulation.
  Interventions: Drug: Dydrogesterone
- Placebo group (Placebo Comparator): Placebo will be given given for two weeks from the next day of the LH surge or hCG induced ovulation.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dydrogesterone — Progesterone
  Other Names: Duphaston
  Arms: Dydrogesterone group
Drug: Placebo — Placebo with appearance similar to Dydrogesterone
  Arms: Placebo group

SUMMARY:
This randomised double-blinded controlled trial aims to compare the live birth rate in natural FET cycles with and without oral dydrogesterone as luteal phase support. The hypothesis is that the use of oral dydrogesterone will increase the live birth rate of natural cycle FET.

DETAILED DESCRIPTION:
Trial design:

Women undergoing FET in the Centre of Assisted Reproduction and Embryology, The University of Hong Kong-Queen Mary Hospital, will be recruited and will be randomized into one of the following two study groups:

Treatment group: Oral dydrogesterone 10mg tds will be given for two weeks from the next day of the LH surge or hCG induced ovulation.

Control group: Placebo will be given given for two weeks from the next day of the LH surge or hCG induced ovulation.

Treatment of subjects

Ovarian stimulation protocol:

All women received ovarian stimulation according to the standard protocol of the Centre. Egg collection is carried out 36 hours after the HCG trigger. One to two early cleaving embryos or blastocysts will be transferred and any excess good quality cleaving embryos or blastocyst will be frozen two to six days after egg collection.

FET cycle:

FET is carried out at least 2 month after the stimulated cycle if the patient fails to get pregnant in the stimulated IVF cycle. Frozen cleaving embryos or blastocysts after thawing are transferred in natural cycles for those women having regular ovulatory cycles. Women are monitored daily from 18 days before the expected date of he next period for pelvic ultrasound assessment of the size of the leading follicle and determination of serum oestradiol (E2) and LH concentrations until the LH surge, which is defined by the LH level being above 20 IU/L and more than double of the average of the LH levels over the past three days. HCG can also be given when the leading follicle reaches 17mm in diameter.

Women will be counseled by a designated research nurse who will explain the purpose of this study when they first attend the clinic for FET. On the day of the hCG trigger or one day after the LH surge, those who consent to join the study will be randomized into one of the two study arms specified in an opaque envelope according to a computer-generated randomization list prepared by a research nurse who is not involved in the present study. Oral dydrogesterone and placebo tablets have the same appearance and will be started one day after the hCG trigger or the LH surge for two weeks.

The transfer is performed on the third day after the LH surge or the fourth day after the hCG trigger for frozen cleaving embryos (on the sixth day after the LH surge or the seventh day after hCG trigger for frozen blastocysts). Again 1-2 cleaving embryos are replaced according to our standard protocol. A urine pregnancy test will be performed 16 days after the FET. In case of pregnancy, the outcome of pregnancy will be traced afterwards and used for analysis. Luteal phase support is not required in those who get pregnant.

ELIGIBILITY:
Inclusion Criteria:

* Age of women <43 years at the time of stimulated IVF
* Replacing early cleavage embryos or blastocysts after thawing

Exclusion Criteria:

* Requiring hormonal replacement cycles
* Use of donor oocytes or embryos
* Undergoing preimplantation genetic testing
* Presence of hydrosalpinx not corrected surgically prior to FET
* Refusal to join the study

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 716 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
live birth rate | 10 months after recruitment
  the number of live birth beyond 22 weeks gestation per transfer cycle

SECONDARY OUTCOMES:
Clinical pregnancy rate | 6 weeks of gestation after recruitment
  the number of women with an intrauterine gestational sac at 5-6 weeks of gestation
Ongoing pregnancy rate | 10 weeks of gestation after recruitment
  the number of intrauterine pregnancies with fetal pulsation beyond 10 gestation per transfer cycle
Pregnancy loss per number of transfer cycles | less than 22 weeks of gestation
  Miscarriage

CONTACTS AND LOCATIONS:
Overall Officials: Ernest HY Ng, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Obstetrics and Gynaecology, Hong Kong, Hong Kong, China